CLINICAL TRIAL: NCT02174406
Title: Clinical Utility of Whole Breast Screening Ultrasound in Patients Undergoing Digital Breast Tomosynthesis
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-119
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Breast Screening
Keywords: Ultrasound; Digital Breast Tomosynthesis; 14-119

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- women scheduled for breast screening: Each patient will have the following:
  * Screening whole breast ultrasound
  * DBT (Full field digital mammography + tomosynthesis views in the CC and MLO projections). The only change in patient management will be the addition of digital breast tomosynthesis views in patients scheduled for FFDM alone. DBT is currently clinically approved and being offered on a voluntary basis to patients scheduled for FFDM.
  Interventions: Procedure: breast ultrasound; Procedure: DBT (Full field digital mammography + tomosynthesis)

INTERVENTIONS:
Procedure: breast ultrasound
Procedure: DBT (Full field digital mammography + tomosynthesis)

SUMMARY:
The purpose of this study is to determine whether ultrasound or Digital breast tomosynthesis (DBT) detects more cancers and to compare the types of cancers detected on ultrasound and DBT.

ELIGIBILITY:
Inclusion Criteria:

* Any women scheduled for screening WBUS and a screening FFDM on the same day or within the following 30 days of each other.

Exclusion Criteria:

* Age < 30 years old
* Male patients
* Patients with any clinical symptoms (palpable mass, nipple discharge, etc)
* Patients with known cancer
* Patients with any breast surgery or biopsy within 90 days prior to the study
* Patients with breast implants
* Patients pregnant or lactating

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women scheduled for a WBUS and a FFDM on the same day or within the following 30 days of each other will be identified by the investigators/research staff at MSKCC clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1494 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
estimate the cancer detection rates | 2 years
  The detection rate of each imaging test is defined as the proportion of patients who are positive on that imaging test who truly have the disease compared to the total number of women screened. A positive imaging test is defined as a test with a recommendation for biopsy (BI-RADS 4 or 5).

CONTACTS AND LOCATIONS:
Overall Officials: Janice Sung, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/